CLINICAL TRIAL: NCT01201798
Title: A Phase 3 Multicenter, Randomized, Double-Masked Study of the Safety and Efficacy of Difluprednate 0.05% Ophthalmic Emulsion Compared to Prednisolone Acetate 1% Ophthalmic Suspension in the Treatment of Endogenous Anterior Uveitis
Brief Title: Safety and Efficacy of Difluprednate 0.05% for the Treatment of Anterior Uveitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-10-034
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Results first posted 2012-11-15 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-10

CONDITIONS: Endogenous Anterior Uveitis
MeSH Terms: interventions — difluprednate; prednisolone acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Durezol (Experimental): Difluprednate 0.05% ophthalmic emulsion, 1 drop in study eye, 4 times a day for 14 days, followed by a 14-day tapering period
  Interventions: Drug: Difluprednate 0.05% ophthalmic emulsion
- Pred Forte (Active Comparator): Prednisolone acetate 1.0% ophthalmic suspension, 1 drop in study eye, 8 times a day for 14 days, followed by a 14-day tapering period
  Interventions: Drug: Prednisolone acetate 1.0% ophthalmic suspension

INTERVENTIONS:
Drug: Difluprednate 0.05% ophthalmic emulsion — 1 drop in study eye, 4 times a day, for 14 days, followed by a 14-day tapering period dependent on the Investigator's determination of adequate response to treatment
  Other Names: Durezol
  Arms: Durezol
Drug: Prednisolone acetate 1.0% ophthalmic suspension — 1 drop in study eye, 8 times a day, for 14 days, followed by a 14-day tapering period dependent on the Investigator's determination of adequate response to treatment
  Other Names: Pred Forte
  Arms: Pred Forte

SUMMARY:
The purpose of this study was to demonstrate that difluprednate 0.05% (Durezol) dosed 4 times daily is noninferior to prednisolone 1% (Pred Forte) dosed 8 times daily for the treatment of endogenous anterior uveitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of endogenous anterior uveitis in at least 1 eye.
* The presence of > 10 cells in the anterior chamber of at least one eye, and a flare score of > 2 in that same eye.
* Age 2 years or older on day of consent.
* Negative urine pregnancy test on Day 0 for females of childbearing potential who are not at least 1 year post-menopausal or surgically sterilized.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Presence of endogenous anterior uveitis diagnosed for > 2 weeks prior to enrollment in the study.
* Presence of intermediate uveitis, posterior uveitis or panuveitis in either eye.
* Instillation of any topical corticosteroid or NSAID in the study eye within 7 days of instillation of study drug.
* History of glaucoma or clinically significant ocular hypertension in the opinion of the Investigator involving an IOP ≥ 21 millimeters mercury in either eye.
* History of steroid-induced elevation of intraocular pressure.
* Any confirmed or suspected active viral, bacterial or fungal keratoconjunctival disease in either eye.
* History of glaucoma or clinically significant ocular hypertension in the opinion of the Investigator involving an intraocular pressure (IOP) > 21 mmHg in either eye.
* Corneal abrasion or ulceration in either eye.
* Pregnancy or lactation.
* Other protocol-defined exclusion criteria may apply.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center, Fort Worth, Texas, United States

REFERENCES:
- [Derived] Sheppard JD, Toyos MM, Kempen JH, Kaur P, Foster CS. Difluprednate 0.05% versus prednisolone acetate 1% for endogenous anterior uveitis: a phase III, multicenter, randomized study. Invest Ophthalmol Vis Sci. 2014 May 6;55(5):2993-3002. doi: 10.1167/iovs.13-12660. PMID 24677110

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 21 US study sites.
Pre-assignment Details: This reporting group includes all randomized subjects: 110. One subject was enrolled but discontinued prior to receiving study medication, with treatment randomization unknown.
Period: Overall Study
Arm/Group | Durezol | Pred Forte
Started | 56 | 54
Completed | 47 | 39
Not Completed | 9 | 15
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 3 | 5
Not completed — Decision Unrelated to an Adverse Event | 1 | 1
Not completed — Noncompliance | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Treatment Failure | 1 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Durezol | Pred Forte | Total
Number analyzed (Participants) | 56 | 54 | 110
Age Continuous [Mean (Standard Deviation); unit: years] | 49.8 (15.20) | 45.5 (18.29) | 47.7 (16.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 60
  Male | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Day 0) in Anterior Chamber Cell Grade at Day 14
Description: Inflammatory cells in the anterior chamber were assessed by the investigator during slit lamp examination and graded on a 5-point scale, with 0 = ≤ 1 cell count; 1 = 2 to 10 cell count; 2 = 11 to 20 cell count; 3 = 21 to 50 cell count; and 4 = > 50 cell count.
Time Frame: Baseline (Day 0), Day 14
Population: Per Protocol: All randomized patients who received at least one dose of the allocated study medication and had no major protocol deviations, including violation of entry criteria, poor compliance, and use of prohibited medications. Last observation carried forward (LOCF) was performed for missing data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Durezol | Pred Forte
Number analyzed (Participants) | 46 | 47
Units on a scale
  Baseline (Day 0) | 2.6 (0.68) | 2.6 (0.68)
  Day 14 | -2.2 (0.96) [-0.53 to 0.09] | -2.0 (1.00)
Statistical Analysis 1: Comparison: Durezol vs Pred Forte; A two-tailed 95% confidence interval was calculated for the difference in change from baseline in anterior chamber cell grade at Day 14 (difluprednate minus prednisolone). The confidence interval was derived from an analysis of covariance (ANCOVA), with investigative site included as a fixed effect to match the stratification used in the randomization process. Treatment and baseline anterior chamber cell grade were also included as fixed effects; Test type: Non-Inferiority or Equivalence — The noninferiority margin was 0.5 units, meaning that the upper limit of the two-tailed 95% confidence interval must have been less than 0.5 to establish noninferiority; ANCOVA; Mean Difference (Net) = -0.22, 95% CI 2-sided [-0.53 to 0.09]

2. Secondary Outcome: Change From Baseline (Day 0) in Anterior Chamber Cell Grade at All Time Points Other Than Day 14
Description: as for outcome 1
Time Frame: Baseline (Day 0), Day 3, Day 7, Day 21, Day 28, Day 35, Day 42
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Durezol | Pred Forte
Number analyzed (Participants) | 46 | 47
Units on a scale
  Baseline (Day 0) | 2.6 (0.68) | 2.6 (0.68)
  Day 3 | -1.1 (0.95) | -1.0 (0.86)
  Day 7 | -1.8 (0.77) | -1.6 (0.85)
  Day 21 | -2.4 (0.98) | -2.1 (0.80)
  Day 28 | -2.3 (0.95) | -2.1 (0.95)
  Day 35 | -2.3 (0.94) | -2.1 (1.04)
  Day 42 | -2.3 (1.00) | -2.1 (1.01)

3. Secondary Outcome: Change From Baseline (Day 0) in Anterior Chamber Flare Grade at All Time Points
Description: Anterior chamber flare (protein escaping from dialated vessels) was assessed by the investigator during slit lamp examination and graded on a 5-point scale, with 0 = none; 1 = mild (trace to clearly noticeable, visible); 2 = moderate; 3 = marked; and 4 = severe.
Time Frame: Baseline (Day 0), Day 3, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Durezol | Pred Forte
Number analyzed (Participants) | 46 | 47
Units on a scale
  Baseline (Day 0) | 2.2 (0.48) | 2.3 (0.54)
  Day 3 | -1.1 (0.83) | -1.2 (1.07)
  Day 7 | -1.6 (0.77) | -1.6 (0.95)
  Day 14 | -2.0 (0.75) | -1.9 (0.91)
  Day 21 | -2.0 (0.77) | -2.0 (0.78)
  Day 28 | -2.0 (0.76) | -2.0 (0.79)
  Day 35 | -2.0 (0.77) | -2.0 (0.83)
  Day 42 | -2.0 (0.77) | -2.0 (0.82)

4. Secondary Outcome: Proportion of Subjects With Anterior Chamber Cell Grade of 0
Description: Inflammatory cells in the anterior chamber were assessed by the investigator during slit lamp examination and graded on a 5-point scale, with 0 = ≤ 1 cell count; 1 = 2 to 10 cell count; 2 = 11 to 20 cell count; 3 = 21 to 50 cell count; and 4 = > 50 cell count. Proportion is reported as percentage of subjects.
Time Frame: Day 3, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | Durezol | Pred Forte
Number analyzed (Participants) | 46 | 47
Percentage of subjects
  Day 3 | 15.2 | 6.4
  Day 7 | 34.8 | 25.5
  Day 14 | 65.2 | 55.3
  Day 21 | 84.8 | 63.8
  Day 28 | 80.4 | 70.2
  Day 35 | 78.3 | 70.2
  Day 42 | 76.1 | 74.5

5. Secondary Outcome: Proportion of Subjects With Anterior Chamber Cell Count of 0
Description: Inflammatory cells in the anterior chamber were assessed by the investigator during slit lamp examination and recorded based on actual cell count. Proportion is reported as a percentage of subjects.
Time Frame: Day 3, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | Durezol | Pred Forte
Number analyzed (Participants) | 46 | 47
Percentage of subjects
  Day 3 | 13.0 | 2.1
  Day 7 | 21.7 | 21.3
  Day 14 | 52.2 | 38.3
  Day 21 | 73.9 | 48.9
  Day 28 | 73.9 | 63.8
  Day 35 | 69.6 | 63.8
  Day 42 | 69.6 | 68.1

6. Secondary Outcome: Proportion of Subjects With Anterior Chamber Cell Count ≤5 and Flare Grade of 0
Description: Inflammatory cells in the anterior chamber were assessed by the investigator during slit lamp examination and recorded based on actual cell count. Anterior chamber flare (protein escaping from dialated vessels) was assessed by the investigator during slit lamp examination and graded on a 5-point scale, with 0 = none; 1 = mild (trace to clearly noticeable, visible); 2 = moderate; 3 = marked; and 4 = severe. Proportion is reported as percentage of subjects.
Time Frame: Day 3, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | Durezol | Pred Forte
Number analyzed (Participants) | 46 | 47
Percentage of subjects
  Day 3 | 13.0 | 14.9
  Day 7 | 41.3 | 40.4
  Day 14 | 78.3 | 61.7
  Day 21 | 82.6 | 76.6
  Day 28 | 80.4 | 76.6
  Day 35 | 82.6 | 76.6
  Day 42 | 80.4 | 78.7

7. Secondary Outcome: Proportion of Subjects With Anterior Chamber Cell Grade ≤1
Description: As assessed by the investigator during slit lamp examination. Anterior chamber cell grade was graded on a 5-point scale, with 0 = no cells; 1 = 1 to 10 cells; 2 = 11 to 20 cells; 3 = 21 to 50 cells; and 4 = more than 50 cells. Proportion is reported as percentage of subjects.
Time Frame: Day 3, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | Durezol | Pred Forte
Number analyzed (Participants) | 46 | 47
Percentage of subjects
  Day 3 | 50.0 | 57.4
  Day 7 | 87.0 | 80.9
  Day 14 | 93.5 | 85.1
  Day 21 | 93.5 | 89.4
  Day 28 | 93.5 | 87.2
  Day 35 | 93.5 | 85.1
  Day 42 | 91.3 | 85.1

8. Secondary Outcome: Proportion of Subjects Who Discontinued Due to Lack of Efficacy
Description: Lack of efficacy was defined as those subjects who discontinued study participation either due to treatment failure or an adverse event with a preferred term of iridocyclitis, iritis, uveitis, or vitritis. Proportion is reported as percentage of subjects.
Time Frame: Time to Event
Population: Per Protocol: All randomized patients who received at least one dose of the allocated study medication and had no major protocol deviations, including violation of entry criteria, poor compliance, and use of prohibited medications.
Measure: Number; unit: Percentage of subjects
Arm/Group | Durezol | Pred Forte
Number analyzed (Participants) | 46 | 47
Percentage of subjects | 0 | 14.9

9. Secondary Outcome: Change From Baseline (Day 0) in Visual Analog Scale (VAS) Total Symptom Score at All Time Points
Description: The following symptoms were each graded by the subject according to a 0-100 visual analog scale (VAS) using a mark on a 100 mm line (0 = absent, 100 = maximal): eye pain, photophobia, blurred vision, and lacrimation. The total symptom score was calculated as the sum of the 4 individual symptom scores.
Time Frame: Baseline (Day 0), Day 3, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Durezol | Pred Forte
Number analyzed (Participants) | 46 | 47
Units on a scale
  Baseline (Day 0) | 186.7 (112.6) | 203.2 (110.8)
  Day 3 | -88.4 (92.55) | -88.4 (92.71)
  Day 7 | -108.2 (114.2) | -123.8 (100.4)
  Day 14 | -133.3 (109.3) | -137.4 (108.8)
  Day 21 | -138.8 (112.7) | -149.5 (108.0)
  Day 28 | -140.1 (111.4) | -152.4 (115.9)
  Day 35 | -143.9 (111.0) | -147.3 (111.3)
  Day 42 | -146.2 (111.7) | -155.5 (112.1)

10. Secondary Outcome: Change From Baseline (Day 0) in Slit-Lamp Total Sign Score at All Visits
Description: The following signs were each graded on a 0 - 3 scale (0 = absent; 1 = mild; 2 = moderate; 3 = severe): posterior synechia, hypopyon, limbal injection, and keratic precipitates. Peripheral synechia was graded by the combined number of clock hours affected (0 = absent; 1 = < 3 hrs; 2 = 3-6 hours; 3 = > 6 hours). The total sign score was calculated as the sum of the 5 individual sign scores, the anterior chamber cell grade and the anterior chamber flare grade. The minimum/best total sign score was 0, and the maximum/worst total sign score was 23.
Time Frame: Baseline (Day 0), Day 3, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Durezol | Pred Forte
Number analyzed (Participants) | 46 | 47
Units on a scale
  Baseline (Day 0) | 7.1 (2.71) | 7.3 (2.87)
  Day 3 | -3.5 (2.71) | -3.6 (2.95)
  Day 7 | -5.2 (2.31) | -5.0 (3.05)
  Day 14 | -6.1 (2.81) | -5.8 (3.34)
  Day 21 | -6.5 (3.07) | -6.2 (3.04)
  Day 28 | -6.4 (2.96) | -6.2 (3.18)
  Day 35 | -6.3 (2.98) | -6.2 (3.34)
  Day 42 | -6.2 (3.21) | -6.3 (3.27)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 9 months, 3 weeks. The safety population consisted of all randomized subjects who received at least 1 dose of the allocated study medication.
Description: Adverse events were obtained as solicited comments from study subjects and observations by study investigator as outlined in study protocol. An adverse event was defined as any untoward medical occurrence in a subject administered a study treatment regardless of causal relationship.
Arm/Group | Durezol | Pred Forte
Serious Adverse Events (participants affected / at risk) | 2/56 | 0/54
Other Adverse Events (participants affected / at risk) | 14/56 | 8/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Durezol (N=56) | Pred Forte (N=54)
Necrotising retinitis (Eye disorders) | 1 | 0 — Non-related
Hypertension (Vascular disorders) | 1 | 0 — Not related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Durezol (N=56) | Pred Forte (N=54)
Iridocyclitis (Eye disorders) | 3 | 2
Punctate keratitis (Eye disorders) | 3 | 0
Intraocular Pressure Increased (Investigations) | 5 | 2
Headache (Nervous system disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Alcon reserves the right of prior review of any publication or presentation of information related to the study.